CLINICAL TRIAL: NCT05009706
Title: Self-care in Older Frail Persons With Heart Failure Intervention (SOPHI). Individualized Physical Exercise, Diet and Symptom Management- A Randomized Controlled Trial.
Brief Title: Self-care in Older Frail Persons With Heart Failure Intervention
Acronym: SOPHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Nana Waldreus, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dnr 2020-00295
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Self Care; Heart Failure; Frailty
Keywords: self care; heart failure; symptom management; exercise; nutrition
MeSH Terms: conditions — Heart Failure; Frailty; Motor Activity | interventions — Self Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Care group (Experimental): Patients who are randomized to the intervention Self Care group will get advice and support on physical excercise, nutrition and symptom management to perform at home for 12 weeks. Once a week, patients will come to the hospital for follow-up and to exercise with a physiotherapist.
  Interventions: Other: Self-care in Older frail Persons with Heart failure Intervention (SOPHI)
- Control group (No Intervention): Patients who are randomized to the Control group will receive ordinary health care (from an outpatient clinic), but will also be encouraged to follow recommendation of 150 minutes/week of moderate physical activity (12 weeks). To compensate for the extra attention received by the intervention group by the advice/support, the patients in the control group will be dialed with a nurse at 3, 6 and 9 weeks to discuss their current activity.

INTERVENTIONS:
Other: Self-care in Older frail Persons with Heart failure Intervention (SOPHI) — Patients who are randomized to the Self Care group will receive oral and written information, advice and support on following activities: excercise (from physiotherapist), nutrition (dietician) and symptom management (nurse), based on patient´s individual needs and abilities. The Self Care group will perform the activities daily at home. Once a week, patients come to the hospital to exercise with the support of a physiotherapist. Once a week or every other week patients will meet (at hospital or by phone) the dietician and nurse to solve possible problems and to follow-up food/nutrition intake and symptoms/symptom management.
  Arms: Self Care group

SUMMARY:
The overall purpose of the randomized controlled study is to evaluate the effects of physical exercise, nutrition and symptom management on physical capacity in older, frail persons with heart failure.

DETAILED DESCRIPTION:
The randomized controlled study will be conducted in order to evaluate the effects of individual needs of physical exercise, nutrition, and symptom management in patients with heart failure who are frail and older. Patients discharged from a geriatric hospital will be recruited and included after informed consent. Two weeks after hospital discharge patients are randomized to intervention or control group. The intervention period is 3 months. With support from a physioterapeut, dietician and a registered nurse, the intervention will be performed in the participants´ home. Once a week participants will come to the hospital for physical exercise led by a physiotherapist. Once a week or every other week participants will meet a dietician and a nurse. Data will be collected at baseline, and 3 and 6 months after baseline. Data consist of e.g. study flow description, number of eligible patients, number of drop-outs, patients sociodemographic- and clinical data, physical function and performance, nutritional status, symptom burden, self-care, appetite, thirst, health-related quality of life. At 12 months after baseline, data will be collected on hospital admissions, reasons for hospital admissions, length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients at geriatric clinic
* Diagnosed with heart failure (independent of Ejection Fraction (EF): both patients with preserved EF or reduced EF can be included
* New York Heart Association functional class II - III
* Clinical frailty level 4-6 (moderate frailty)
* Discharge from hospital to home

Exclusion Criteria:

* New York Heart Associacion functional class I or IV
* Clinical frailty level 1-3 (no/mild frailty) and 7-9 (severe frailty)
* The patient is unable to perform gait tests due to visual (see a TV screen at a 3 meter distance), cognitive (assessed by nurse or doctor) or motor impairment (the patient should be able to stand up from sitting and have the ability to walk with or without a walker or other walking aid).
* The patient is unable to follow instructions (assessed by nurse or doctor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in physical performance | 3 months
  The "Short Physical Performance Battery" is composed of "standing balance", "gait speed", and "timed repeated chair rise". The total score range from minimum 0 to maximum 12, with higher scores indicating better physical performance.

SECONDARY OUTCOMES:
Symptom burden | Baseline, 3 and 6 months
  Assessed by the questionnaire titled "The Memorial Symptom Assessment Scale- Heart Failure", that evaluates symptoms experienced by the patient in the last week (a total of 36 symptoms, for example pain, nausea, tiredness). A score of 0 is given to a symptom if it is absent. If the symptom is present, it is rated using a four-point rating scale (1-4) for frequency and severity, and a five-point rating scale (0-4) for distress of the symptom with higher scores indicating greater frequency, more severity and higher distress. For each symptom, the average of the frequency, severity and distress will be calculated to produce the outcome symptom burden (total scores ranging from minimum 0 to maximum 4, with higher scores indicating greater symptom burden).
Health related quality of life | Baseline, 3 and 6 months
  Assessed with the Euroqol questionnaire titled "The EQ-5D". It comprises five questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Answer options are no problems (score 1), moderate problems (score 2), severe/extreme problems (score 3). The results are converted into a single index value (minimum value 0 to maximum value 1). Higher value indicate better health related quality of life
Aerobic capacity/endurance | Baseline, 3 and 6 months
  Assessed with the 6-minute walk test, the distance in meters covered over a time of 6 minutes
Frailty | Baseline, 3 and 6 months
  Assessed by the scale titled "Clinical Frailty Scale". From the minimum value 1 (patient is very fit) to the maximum value 9 (terminally ill). Higher score indicates more frailty
Perceived physical effort | Baseline, 3 and 6 months
  Assessed with the scale titled "Borg Category Ratio-10 Scale" of perceived exertion.
  The minimum value is 0 (nothing at all) to the maximum value 10 (extremely strong or maximal). Higher value indicate worse physical effort
Hand strength | Baseline, 3 and 6 months
  Assessed with the hand-gripdynamometer (JAMAR)
Hospital readmissions | 12 months
  The number of hospital readmissions during a 12 month period will be retrieved from the patients medical record
Lower body strength | Baseline, 3 and 6 months
  Sit to stand test measure the number of uprising from a chair during 30 seconds
Nutrition status | Baseline, 3 and 6 months
  Assessed by the "Mini Nutritional Assessment" screening. The total score range from minimum 0 to maximum 14. Higher scores indicate better nutrition status
Inflammation marker | Baseline, 3 and 6 months
  Plasma C-reactive protein (mg/L), reference interval value below 3 mg/L. Higher value indicate inflammation in the body
Sarcopenia | Baseline, 3 and 6 months
  Measured by the criteria of European Working Group on Sarcopenia in Older People's

OTHER OUTCOMES:
Objective physical activity | Baseline, 3 and 6 months
  Measured with a non-invasive miniature electronic logger during 4-5 days per time frame
Subjective physical activity | Baseline, 3 and 6 months
  Assessed by the instrument titled "International Physical Activity Questionnaire" (IPAQ). Measure the minutes of physical activity during a day.
Experiences of patients | 3 months
  A qualitative interview will be used to collect data on patient´s experiences of the intervention
Self-care | Baseline, 3 and 6 months
  Assessed with the questionnaire titled "Self-care of chronic illness inventory" (30 questions).
  Minimum score is 28 and maximum score is 150. Higher score indicate better self care
Appetite | Baseline, 3 and 6 months
  Assessed with the questionnaire titled "The Council on Nutrition Appetite Questionnaire" (8 questions)Failure".
  Minimum score is 8 and maximum score is 40. Higher score indicate better appetite
Thirst distress | Baseline, 3 and 6 months
  Assessed with the questionnaire titled "Thirst Distress Scale for patients with Heart Failure" (8 questions) Minimum score is 8 and maximum score is 40. Higher score indicate higher thirst distress

CONTACTS AND LOCATIONS:
Overall Officials: Nana Waldréus, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Universitetssjukhuset, Tema Inflammation och Åldrande, Huddinge, Sweden